CLINICAL TRIAL: NCT01860170
Title: A Phase I Trial of Post-Transplant Bortezomib and High Dose Cyclophosphamide as Graft-Versus-Host Disease (GVHD) Prophylaxis After Reduced-Intensity Allogeneic Hematopoietic Stem Cell Transplantation (AHSCT)
Brief Title: Post-Transplant Bortezomib and High Dose Cyclophosphamide as Graft-Versus-Host Disease (GVHD) Prophylaxis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Corewell Health West (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2013-083
Record Dates: First submitted 2013-05-14; First posted 2013-05-22 (Estimated); Results first posted 2017-05-17 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Hematological Malignancy
Keywords: Blood and Marrow Transplant (BMT); MRD; MUD; GVHD
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Bortezomib; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1-Bortezomib (Velcade®) (Active Comparator): Bortezomib (Velcade®) 0.7 mg/m2 rapid IV push on days 0 (at least 6 hours after transplant) and +3.
  Interventions: Drug: Cohort 1-Bortezomib (Velcade ®)
- Cohort 2-Bortezomib (Velcade®) (Active Comparator): Bortezomib (Velcade®) 1 mg/ m2 rapid IV push on days 0 (at least 6 hours after transplant) and +3.
  Interventions: Drug: Cohort 2-Bortezomib (Velcade ®)
- Cohort 3-Bortezomib (Velcade®) (Active Comparator): Bortezomib (Velcade®) 1.3 mg/m2 rapid IV push on days 0 (at least 6 hours after transplant) and +3.
  Interventions: Drug: Cohort 3-Bortezomib (Velcade ®)

INTERVENTIONS:
Drug: Cohort 1-Bortezomib (Velcade ®) — Conditioning Regimen: Fludarabine 30 mg/m2 on days -7, -6, -5, -4, -3 and -2; Busulfan 0.8 mg/kg, every 6 hours on days -3 and -2; Patients with matched unrelated donor also receive rATG (Thymoglobulin ®) 2 mg/kg on days -4, -3, -2 and -1.
  Cyclophosphamide 50 mg/kg, in 500 mL NS over 2 hours on days +3 and +4. Concomitant hydration with NS with 20 mEq/L at 250 mL/hr starting 4 hours before and continuing until 24 hours after the second dose is given. Furosemide on as needed basis to maintain fluid balance is also given. It is important to avoid administration of any immunosuppressive drugs include steroids after day 0.
  Bortezomib 0.7 mg/m2 rapid IV push on days 0 (at least 6 hours after transplant) and +3.
  Other Names: Cyclophosphamide (Cytoxan ®); Bortezomib (Velcade ®)
  Arms: Cohort 1-Bortezomib (Velcade®)
Drug: Cohort 2-Bortezomib (Velcade ®) — Conditioning Regimen: Fludarabine 30 mg/m2 on days -7, -6, -5, -4, -3 and -2; Busulfan 0.8 mg/kg, every 6 hours on days -3 and -2; Patients with matched unrelated donor also receive rATG (Thymoglobulin ®) 2 mg/kg on days -4, -3, -2 and -1.
  Cyclophosphamide 50 mg/kg, in 500 mL NS over 2 hours on days +3 and +4. Concomitant hydration with NS with 20 mEq/L at 250 mL/hr starting 4 hours before and continuing until 24 hours after the second dose is given. Furosemide on as needed basis to maintain fluid balance is also given. It is important to avoid administration of any immunosuppressive drugs include steroids after day 0.
  Bortezomib 1 mg/ m2 rapid IV push on days 0 (at least 6 hours after transplant) and +3.
  Other Names: Cyclophosphamide (Cytoxan ®); Bortezomib (Velcade ®)
  Arms: Cohort 2-Bortezomib (Velcade®)
Drug: Cohort 3-Bortezomib (Velcade ®) — Conditioning Regimen: Fludarabine 30 mg/m2 on days -7, -6, -5, -4, -3 and -2; Busulfan 0.8 mg/kg, every 6 hours on days -3 and -2; Patients with matched unrelated donor also receive rATG (Thymoglobulin ®) 2 mg/kg on days -4, -3, -2 and -1.
  Cyclophosphamide 50 mg/kg, in 500 mL NS over 2 hours on days +3 and +4. Concomitant hydration with NS with 20 mEq/L at 250 mL/hr starting 4 hours before and continuing until 24 hours after the second dose is given. Furosemide on as needed basis to maintain fluid balance is also given. It is important to avoid administration of any immunosuppressive drugs include steroids after day 0.
  Bortezomib 1.3 mg/m2 rapid IV push on days 0 (at least 6 hours after transplant) and +3.
  Other Names: Cyclophosphamide (Cytoxan ®); Bortezomib (Velcade ®)
  Arms: Cohort 3-Bortezomib (Velcade®)

SUMMARY:
The purpose of this study is to determine if Bortezomib, known commercially as Velcade is safe and tolerated at different dose levels (amounts) with high dose Cyclophosphamide to be used as graft versus host disease prevention after reduced-intensity allogeneic hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
It is hypothesized that the administration of an early and short course cyclophosphamide and bortezomib after allogeneic hematopoietic stem cell transplantationin in the setting of matched related or unrelated donor transplantation using a standard reduced-intensity conditioning regimen is feasible.

The study is a phase I study. The primary objective of the study is to determine the feasibility and safety of increasing doses of bortezomib administered post-transplant in conjunction with fixed high dose cyclophosphamide, also administered post-transplant in the setting of reduced-intensity allogeneic hematopoietic stem cell transplant, as GVHD prophylaxis strategy. Eligible patients will receive a conditioning regimen based on a combination of fludarabine and busulfan with or without rATG.

ELIGIBILITY:
Inclusion Criteria

1. 8 out of 8 matched related or unrelated donor
2. Age > 18 years
3. Good performance status with a Karnofsky score >/= to 70%
4. No evidence of progressive bacterial, viral or fungal infection despite adequate treatment
5. Creatinine clearance > 40 mL/min/1.72m2
6. Total bilirubin < 1.5 and ALT and AST < 2 times the upper limit of normal
7. Cardiac ejection fraction > 40%
8. DLCO > 50%
9. Negative pregnancy test
10. Negative HIV serology
11. Able to provide informed consent
12. Female subject is either postmenopausal for at least 1 year before the screening visit, is surgically sterilized or if they are of childbearing potential, agree to practice 2 effective methods of contraception from the time of signing the informed consent form through 30 days after the last dose of bortezomib, or agree to completely abstain from heterosexual intercourse.
13. Male subjects, even if surgically sterilized (ie, status postvasectomy) must agree to 1 of the following: practice effective barrier contraception during the entire study treatment period and through a minimum of 30 days after the last dose of study drug, or completely abstain from heterosexual intercourse.

Exclusion Criteria:

1. Age <18 years
2. Poor performance status (<70%)
3. Active infections
4. Abnormal creatinine clearance <40ml/min
5. Elevated bilirubin >1.5 and ALT and AST .2 times the upper limit of normal
6. Poor ejection fraction <40%
7. DLCO <50%
8. Pregnant female.
9. HIV positive
10. Inability to provide informed consent
11. Patient has >/= Grade 2 peripheral neuropathy
12. Patient had myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at screening must be documented by the investigator as not medically relevant.
13. Patient has hypersensitivity to bortezomib, boron, or mannitol.
14. Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
15. Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy.
16. Participation in clinical trials with other investigational agents not included in this trial, within 14 days of the start of this trial and throughout the duration of this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A. Samer Al-Homsi, MD, Principal Investigator — Corewell Health West
Locations (1):
- Spectrum Health, Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1-Bortezomib (Velcade®): Bortezomib (Velcade®) 0.7 mg/m2 rapid IV push on days 0 (at least 6 hours after transplant) and +3.
  Cohort 1-Bortezomib (Velcade ®): Conditioning Regimen: Fludarabine 30 mg/m2 on days -7, -6, -5, -4, -3 and -2; Busulfan 0.8 mg/kg, every 6 hours on days -3 and -2; Patients with matched unrelated donor also receive rATG (Thymoglobulin ®) 2 mg/kg on days -4, -3, -2 and -1.
  Cyclophosphamide 50 mg/kg, in 500 mL NS over 2 hours on days +3 and +4. Concomitant hydration with NS with 20 mEq/L at 250 mL/hr starting 4 hours before and continuing until 24 hours after the second dose is given. Furosemide on as needed basis to maintain fluid balance is also given. It is important to avoid administration of any immunosuppressive drugs include steroids after day 0.
  Bortezomib 0.7 mg/m2 rapid IV push on days 0 (at least 6 hours after transplant) and +3.
- Cohort 2-Bortezomib (Velcade®): Bortezomib (Velcade®) 1 mg/ m2 rapid IV push on days 0 (at least 6 hours after transplant) and +3.
  Cohort 2-Bortezomib (Velcade ®): Conditioning Regimen: Fludarabine 30 mg/m2 on days -7, -6, -5, -4, -3 and -2; Busulfan 0.8 mg/kg, every 6 hours on days -3 and -2; Patients with matched unrelated donor also receive rATG (Thymoglobulin ®) 2 mg/kg on days -4, -3, -2 and -1.
  Cyclophosphamide 50 mg/kg, in 500 mL NS over 2 hours on days +3 and +4. Concomitant hydration with NS with 20 mEq/L at 250 mL/hr starting 4 hours before and continuing until 24 hours after the second dose is given. Furosemide on as needed basis to maintain fluid balance is also given. It is important to avoid administration of any immunosuppressive drugs include steroids after day 0.
  Bortezomib 1 mg/ m2 rapid IV push on days 0 (at least 6 hours after transplant) and +3.
- Cohort 3-Bortezomib (Velcade®): Bortezomib (Velcade®) 1.3 mg/m2 rapid IV push on days 0 (at least 6 hours after transplant) and +3.
  Cohort 3-Bortezomib (Velcade ®): Conditioning Regimen: Fludarabine 30 mg/m2 on days -7, -6, -5, -4, -3 and -2; Busulfan 0.8 mg/kg, every 6 hours on days -3 and -2; Patients with matched unrelated donor also receive rATG (Thymoglobulin ®) 2 mg/kg on days -4, -3, -2 and -1.
  Cyclophosphamide 50 mg/kg, in 500 mL NS over 2 hours on days +3 and +4. Concomitant hydration with NS with 20 mEq/L at 250 mL/hr starting 4 hours before and continuing until 24 hours after the second dose is given. Furosemide on as needed basis to maintain fluid balance is also given. It is important to avoid administration of any immunosuppressive drugs include steroids after day 0.
  Bortezomib 1.3 mg/m2 rapid IV push on days 0 (at least 6 hours after transplant) and +3.
Period: Overall Study
Arm/Group | Cohort 1-Bortezomib (Velcade®) | Cohort 2-Bortezomib (Velcade®) | Cohort 3-Bortezomib (Velcade®)
Started | 3 | 3 | 22
Completed | 3 | 3 | 22
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1-Bortezomib (Velcade®) | Cohort 2-Bortezomib (Velcade®) | Cohort 3-Bortezomib (Velcade®) | Total
Number analyzed (Participants) | 3 | 3 | 22 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 17 | 22
  >=65 years | 1 | 0 | 5 | 6
Age, Continuous [Mean (Full Range); unit: years] | 60.3 [56 to 65] | 56 [47 to 62] | 56.6 [37 to 70] | 56.9 [37 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 7 | 12
  Male | 0 | 1 | 15 | 16
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 22 | 28

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicity
Description: Grade 3 non-hematologic Common Toxicity Criteria toxicity directly related to bortezomib (such as peripheral neuropathy) or Grade 2 or > hepatic bilirubin Common Toxicity Criteria Graft failure
Time Frame: Assessed daily (while inpatient) through clinical and laboratory examination up to 90 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1-Bortezomib (Velcade®) | Cohort 2-Bortezomib (Velcade®) | Cohort 3-Bortezomib (Velcade®)
Number analyzed (Participants) | 3 | 3 | 22
Participants | 0 | 0 | 0

2. Secondary Outcome: Engraftment
Description: Neutrophil engraftment is defined as achieving an absolute neutrophil count (ANC) > 0.5 109/L for 3 consecutive measurements on different days. The first of the 3 days will be considered the day of neutrophil engraftment.
  Platelet engraftment is defined as platelet count > 20 109/L for 3 consecutive measurements over at least 3 days. The first of the 3 days will be considered the day of platelet engraftment.
  In this study, graft failure is defined as lack of achieving neutrophil engraftment by day 22 and donor chimerism > 50% by day 45.
Time Frame: Assessed daily by laboratory evaluation until engraftment or up to 90 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1-Bortezomib (Velcade®) | Cohort 2-Bortezomib (Velcade®) | Cohort 3-Bortezomib (Velcade®)
Number analyzed (Participants) | 3 | 3 | 22
Participants
  Neutrophil Engraftment | 3 | 3 | 22
  Platelet Engraftment | 3 | 1 | 22
  Graft Failure | 0 | 0 | 0

3. Other Pre Specified Outcome: GVHD
Description: aGVHD onset at a certain grade will be used to calculate the cumulative incidence for that grade (e.g., onset of grade 70 post-transplant , time to grade III is 70 days). This end point will be evaluated through day 150 post-transplant. The diagnosis of aGVHD is based on clinical and pathological evaluation by the treating physician.
  The first day of cGVHD will be used to calculate the cumulative incidence of cGVHD. The diagnosis of cGVHD is based on clinical and pathological evaluation by the treating physician.
Time Frame: Assessed routinely by clinical and pathological evaluation. Acute GVHD will be assessed up to day 150 post-transplant. Chronic GVHD will be assess up to 2 years post-transplant.
Measure: Number; unit: participants
Arm/Group | Cohort 1-Bortezomib (Velcade®) | Cohort 2-Bortezomib (Velcade®) | Cohort 3-Bortezomib (Velcade®)
Number analyzed (Participants) | 3 | 3 | 22
participants
  Acute GvHD Grade II-IV | 0 | 0 | 10
  Acute GvHD Grade III-IV | 0 | 0 | 3
  Chronic GvHD | 1 | 1 | 5

ADVERSE EVENTS:
Arm/Group | Cohort 1-Bortezomib (Velcade®) | Cohort 2-Bortezomib (Velcade®) | Cohort 3-Bortezomib (Velcade®)
All-Cause Mortality (participants affected / at risk) | 0/3 | 3/3 | 10/22
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/3 | 6/22
Other Adverse Events (participants affected / at risk) | 1/3 | 2/3 | 19/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1-Bortezomib (Velcade®) (N=3) | Cohort 2-Bortezomib (Velcade®) (N=3) | Cohort 3-Bortezomib (Velcade®) (N=22)
Progressive multifocal leukoencephalopathy (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hypovolemic shock (General disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Fever (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
HSV (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Syncope related to anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1-Bortezomib (Velcade®) (N=3) | Cohort 2-Bortezomib (Velcade®) (N=3) | Cohort 3-Bortezomib (Velcade®) (N=22)
Cytomegalovirus (Infections and infestations) | 1 (1) | 1 (1) | 14 (14)
Epstein-Barr virus (Infections and infestations) | 0 (0) | 1 (1) | 9 (9)
Respiratory syncytial virus (Infections and infestations) | 0 (0) | 1 (1) | 3 (3)
BK virus (Infections and infestations) | 0 (0) | 0 (0) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes